CLINICAL TRIAL: NCT07287358
Title: CPPopt Guided Therapy: Assessment of Target Effectiveness - II
Brief Title: Optimal Cerebral Perfusion Pressure Guided Therapy: Assessment of Target Effectiveness - II
Acronym: Cogitate II
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Medisch Spectrum Twente (Other); Radboud University Medical Center (Other); Medical Center Haaglanden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL-010951
Record Dates: First submitted 2025-11-20; First posted 2025-12-17 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Traumatic Brain Injury; Severe Traumatic Brain Injury; Intracranial Pressure; Cerebral Perfusion Pressure
Keywords: CPPopt; optimal cerebral perfusion pressure; pressure reactivity index; PRx; Intracranial pressure; cerebral perfusion pressure; traumatic brain injury; severe traumatic brain injury; cogitate; cogitate-II
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPPopt treatment (Experimental): The CPPopt treatment group will receive management according to the Brain Trauma Foundation (BTF) guidelines, except for the targeted cerebral perfusion pressure. Here, the calculated "optimal cerebral perfusion pressure (CPPopt)" will be targeted, with updated CPPopt targets every 4 hours.
  Interventions: Other: Optimal cerebral perfusion pressure
- Control group (No Intervention): The intervention group will receive standard brain trauma management according to the Brain Trauma Foundation (BTF) guidelines, including the standard cerebral perfusion pressure target of 60-70 mmHg.

INTERVENTIONS:
Other: Optimal cerebral perfusion pressure — The intervention group will receive CPPopt guided management with updated CPPopt targets every 4 hours. All other parameters will be handled according to Brain Trauma Foundation (BTF) guidelines.
  Other Names: CPPopt
  Arms: CPPopt treatment

SUMMARY:
After severe traumatic brain injury, adequate blood flow to the brain is essential for recovery. This depends on arterial blood pressure, yet intensive care units apply fixed targets to all patients - treating every brain and patient the same. This study aims to change that. With new technology, 'optimal' blood pressure can be determined for each individual brain and treatment can be tailored accordingly. This personalized approach to neurocritical care has never been tested in a randomized controlled study before. If effective in showing reduced brain damage biomarkers, it will fundamentally transform brain injury treatment and dramatically improve recovery outcomes for patients worldwide.

DETAILED DESCRIPTION:
Rationale: In traumatic brain injury patients with intracranial pressure monitoring (TBIicp), individual optimal cerebral perfusion pressure (also called CPPopt) can be determined based on continuous cerebral autoregulation information. In a 2021 study, CPPopt guided management has been demonstrated to be both feasible and safe in clinical practice. This study was performed in 4 European countries and coordinated by the Intensive care department in Maastricht. CPPopt guided management aims to minimize harm from global or regional hypo- or hyperperfusion of the injured brain compared to the classical treatment. Classical treatment maintains cerebral perfusion pressure (CPP) at a fixed, pre-determined range of 60-70 mmHg in all patients during the entire period the intracranial pressure (ICP) is monitored. CPP is calculated as the arterial blood pressure (ABP) minus the ICP. CPP targets are obtained by manipulating ICP (if elevated) or ABP. Observational data suggests that management of CPP above CPPopt is associated with severe disability, and below CPPopt with mortality. However, there is no prospective evidence to support the effectiviness of CPPopt guided management and its effect on clinical outcome in severe TBIicp patients.

Objective: To determine whether individualized CPPopt guided management reduces secondary brain injury in patients with severe traumatic brain injury requiring intracranial pressure monitoring, as reflected by lower concentrations of brain injury-related biomarkers during the first five days of intensive care unit (ICU) admission, compared with standard guideline-based CPP management.

Study design: Multicenter, randomized, controlled trial to test the effectiviness of CPPopt guided management in 4 Dutch hospitals.

Study population: Adult patients with severe traumatic brain injury and intracranial pressure monitoring (TBIicp). 60 patients will be included in a 2 year period.

Intervention: The intervention group will receive CPPopt guided management with updated CPPopt targets every 4 hours, whereas the control group will receive standard of care CPP management formulated as a CPP between 60-70 mmHg according to Brain Trauma Foundation (BTF) guideline.

Main study parameters/endpoints:

The primary outcome of this effectiviness study will be the cumulative release of blood biomarker Glial Fibrillary Acidic Protein (GFAP) over the first five days of ICU admission, quantified as the area under the curve (AUC) in both groups. GFAP is selected because its relatively short half-life makes it particularly sensitive to secondary brain injury, as increases or sustained elevations reflect ongoing damage rather than the initial trauma. In the present study, the hypothesis is that patients managed with CPPopt-guided therapy will show lower cumulative GFAP release over the first five days of ICU admission compared to patients receiving standard guideline-based CPP management. A lower cumulative GFAP level would indicate less secondary neuronal injury during the critical early phase after TBI.

Secondary study parameters are

1. The cumulative release of five additional brain injury biomarkers: Neuron Specific Enolase (NSE), Ubiquitin C-terminal hydrolase L1 (UCH-L1), S100 calcium-binding protein B (S100B), Tau, and Neurofilament light chain (NfL). These biomarkers reflect damage in different brain cell types and structures, and their varying half-lives allow tracking of brain injury dynamics over time. Blood for all biomarker analyses will be stored locally at -80°C until the study end, and then sent in batch to an ISO 15189 accredited laboratory in the Medisch Spectrum Twente for analysis.
2. Cerebral swelling (edema) and hematoma progression will be quantified by comparing brain CT scans obtained at admission with follow-up scans within the first five days of ICU admission (performed when clinically indicated). These imaging data will be used to evaluate the radiological progression of secondary brain injury.
3. Daily Therapy Intensity Level (TIL) score during the first five days on ICU to test whether the intervention reduces the need for aggressive treatment of increased ICP. The TIL score provides a standardized quantitative measure of the therapeutic burden required to manage ICP, with higher scores indicating more intensive treatment. A lower mean daily TIL score in the intervention group would therefore suggest improved ICP stability and potentially less secondary brain injury. A change in daily TIL score of > 3 is representative of a clinically significant effect.
4. Mean daily Pressure Reactivity Index (PRx) values will be calculated as a global measure of cerebral autoregulation. PRx is defined as the moving correlation coefficient between slow waves of ABP and ICP, with more positive values indicating impaired autoregulation. This parameter will be used to assess whether the degree of cerebral autoregulatory function differs between the CPPopt guided intervention group and the standard CPP management (control) group over the first five days of ICU admission.
5. Frequency and cumulative duration of CPP excursions outside the predefined safety limits (CPP between 50 mmHg and 100 mmHg) during the first five days will be recorded for each patient. These data will be used to evaluate the safety of CPPopt guided management compared to standard care, by quantifying both the number and total time of CPP deviations beyond clinically acceptable thresholds.
6. Glasgow Coma Score at ICU discharge will be recorded as an early indicator of patient outcome.
7. ICU mortality will also be recorded as an early indicator of patient outcome. (8) Non-invasive near-infrared spectroscopy (NIRS) values will be recorded using bifrontal sensors to estimate cerebral oxygenation. NIRS provides a non-invasive measure of cerebral perfusion, as changes in cerebral oxygenation correlate with changes in cerebral blood flow. In addition, the correlation between slow waves of NIRS and ABP can be used in selected patients to estimate cerebral autoregulation and to derive non-invasive CPPopt targets. As part of exploratory research, the agreement between non-invasive NIRS-based CPPopt and invasive ICP-based CPPopt will be evaluated in the intervention group. If validated, non-invasive CPPopt-guided management could potentially extend autoregulation-guided therapy to a broader patient population.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years old)
* Severe TBI requiring ICP-directed therapy for at least 24 hrs on the assessment of the recruiting intensive care team and/or attending neurosurgeon
* Start randomization within 24 hrs after ICU admission.

Exclusion Criteria:

* Known pregnancy
* Moribund at presentation (e.g. bilaterally absent pupillary responses)
* Patients with a primary decompressive craniectomy
* Failure to get final written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-15 (Estimated)

PRIMARY OUTCOMES:
Cumulative concentration of blood biomarker Glial Fibrillary Acidic Protein (GFAP) during first 5 days of ICU admission | The first 5 days of ICU admission
  The cumulative release of blood biomarker Glial Fibrillary Acidic Protein (GFAP) over the first five days of ICU admission, quantified as the area under the curve (AUC) in both groups

SECONDARY OUTCOMES:
Cumulative concentrations of biomarkers NSE, UCH-L1, S100B, Tau and NfL during first 5 days of ICU admission | the first 5 days of ICU admission
  The cumulative release of five additional brain injury biomarkers: Neuron Specific Enolase (NSE), Ubiquitin C-terminal hydrolase L1 (UCH-L1), S100 calcium-binding protein B (S100B), Tau, and Neu-rofilament light chain (NfL) over the first 5 days of ICU admission.
Progression of cerebral edema on CT imaging based on size of hypodense regions in sequential CT scans | first five days of ICU admission
  Cerebral edema progression will be quantified by comparing brain CT scans obtained at admission with follow-up scans within the first five days of ICU admission (performed when clinically indicated).
Daily Therapy Intensity Level (TIL) score | first five days on ICU
  Daily intracranial hypertenstion Therapy Intensity Level (TIL) score during the first five days on ICU to test whether our intervention reduces the need for aggressive treatment of increased ICP.
  Individual ICP-targeting therapies were assigned a score based on published estimates of their relative efficacy and risks of morbidity. The TIL includes eight ICP-treatment modalities, termed items. The maximum score is 38, with a higher score indicating that a patient is receiving more complex, aggressive, or frequent treatments.
Mean daily Pressure Reactivity Index (PRx) values | First 5 days on ICU
  Mean daily Pressure Reactivity Index (PRx) values will be calculated as a global measure of cerebral autoregulation. PRx is defined as the moving correlation coefficient between slow waves of ABP and ICP, with more positive values indicating impaired autoregulation.
Frequency and duration of CPP outside safety limits (50-100 mmHg) | First 5 days on ICU
  Frequency and cumulative duration of CPP excursions outside the predefined safety limits (CPP between 50 mmHg and 100 mmHg) during the first five days will be recorded for each patient. These data will be used to evaluate the safety of CPPopt guided management compared to standard care, by quantifying both the number and total time of CPP deviations beyond clinically acceptable thresholds.
Glasgow Coma Score at the moment of intensive care unit discharge | At the moment a patient is discharged from ICU, assessed up to 2 months after ICU admission
  Glasgow Coma Score at ICU discharge will be recorded as an early indicator of patient outcome.
  The Glasgow Coma Scale (GCS) is a clinical diagnostic tool widely used since the 1970s to roughly assess an injured person's level of brain damage. The GCS diagnosis is based on a patient's ability to respond and interact with three kinds of behaviour: eye movements, speech, and other body motions. A GCS score can range from 3 (completely unresponsive) to 15 (responsive). The higher the value, the better the neurological state.
ICU mortality at the moment of ICU discharge | At time of death, or if survival: at the moment the patient is discharged from ICU, assessed up to 2 months after ICU admission
  ICU mortality will also be recorded as an early indicator of patient outcome. Patients dying will be registered as "dead", patients who are alive at ICU discharge will be registered as "survival".
Non-invasive near-infrared spectroscopy (NIRS) values | First 5 days on ICU
  Non-invasive near-infrared spectroscopy (NIRS) values will be recorded using bifrontal sensors to estimate cerebral oxygenation. NIRS provides a non-invasive measure of cerebral perfusion, as changes in cerebral oxygenation correlate with changes in cerebral blood flow
Progression of cerebral hematoma on CT imaging based on size of hyperdense regions in sequential CT scans | First 5 days of ICU admission
  Cerebral hematoma progression will be quantified by comparing brain CT scans obtained at admission with follow-up scans within the first five days of ICU admission (performed when clinically indicated).

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - Medisch Spectrum Twente, Enschede
  - Maastricht Universitair Medisch Centrum+, Maastricht
  - Radboud University Medical Center, Nijmegen
  - Haaglanden Medisch Centrum, The Hague

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Weiss M, Meyfroidt G, Aries MJH. Individualized cerebral perfusion pressure in acute neurological injury: are we ready for clinical use? Curr Opin Crit Care. 2022 Apr 1;28(2):123-129. doi: 10.1097/MCC.0000000000000919. PMID 35058408
- [Background] Beqiri E, Tas J, Czosnyka M, van Kaam RCR, Donnelly J, Haeren RH, van der Horst ICC, Hutchinson PJ, van Kuijk SMJ, Liberti AL, Menon DK, Hoedemaekers CWE, Depreitere B, Meyfroidt G, Ercole A, Aries MJH, Smielewski P. Does Targeting CPP at CPPopt Actually Improve Cerebrovascular Reactivity? A Secondary Analysis of the COGiTATE Randomized Controlled Trial. Neurocrit Care. 2025 Jun;42(3):937-944. doi: 10.1007/s12028-024-02168-y. Epub 2024 Dec 2. PMID 39623160
- [Background] Tas J, Beqiri E, van Kaam RC, Czosnyka M, Donnelly J, Haeren RH, van der Horst ICC, Hutchinson PJ, van Kuijk SMJ, Liberti AL, Menon DK, Hoedemaekers CWE, Depreitere B, Smielewski P, Meyfroidt G, Ercole A, Aries MJH. Targeting Autoregulation-Guided Cerebral Perfusion Pressure after Traumatic Brain Injury (COGiTATE): A Feasibility Randomized Controlled Clinical Trial. J Neurotrauma. 2021 Oct 15;38(20):2790-2800. doi: 10.1089/neu.2021.0197. Epub 2021 Aug 16. PMID 34407385